CLINICAL TRIAL: NCT05762263
Title: The Effect of Flexitarian, Time-restricted Eating on Cardiometabolic Traits in Normal Weight, Young Men: a Factorial Randomized Controlled Trial (FlexiFast Study)
Brief Title: The Effect of Flexitarian, Time-restricted Eating on Cardiometabolic Traits in Normal Weight, Young Men
Acronym: FlexiFast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Marta Lonnie, Principal Investigator, University of Warmia and Mazury in Olsztyn
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2021/41/N/NZ9/01129
Record Dates: First submitted 2022-12-21; First posted 2023-03-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cardiometabolic Syndrome; Glucose Metabolism Disorders; Blood Pressure; Lipid Metabolism Disorders
MeSH Terms: conditions — Metabolic Syndrome; Glucose Metabolism Disorders; Lipid Metabolism Disorders | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Habitual diet - healthy eating guidelines provided for ethical reasons, no restrictions on the time of eating
- Flexitarian diet group (Experimental): Flexitarian diet (FD) will be based on planetary diet recommendations (predominantly plants; pulses and legumes as protein sources, meat and poultry consumed occasionally). Ways to facilitate this diet will be presented in the booklet prepared for them by the PI and a dietitian.
  Interventions: Behavioral: Dietary
- Time-restricted eating group (Experimental): Time restricted eating (TRE) with 6 hour eating window - start and end hour to be an individual choice (some may prefer to consume their meals within an early window, e.g. 10am-4pm, some may prefer to consume their meals later in the day, e.g. 12:00-6pm). However, participants will be asked to be fairly consistent with their choice of their timing of eating hours. During fasting only water will be permitted;
  Interventions: Behavioral: Dietary
- Flexitarian diet & time-restricted eating group (Experimental): Treatment TRE and FD combined.
  Interventions: Behavioral: Dietary

INTERVENTIONS:
Behavioral: Dietary — Depending on the allocation arm, participants will be advised to follow a particular dietary plan (either flexitarian eating, time-restricted eating or both combined).
  Arms: Flexitarian diet & time-restricted eating group; Flexitarian diet group; Time-restricted eating group

SUMMARY:
The goal of this factorial randomized controlled trial is to find out whether time-restricted eating and flexitarian diet (on its own and combined) can improve cardiometabolic health markers in normal weight, young men with metabolic abnormalities?

Participants will be assigned to four groups: control, flexitarian, time-restricted eating and time-restricted eating + flexitarian. Investigators will look for men with elevated fasting blood glucose or blood lipids level or blood pressure and with normal body weight and waistline. Participants from the flexitarian group will be asked to follow a diet that has been carefully designed for them by the PI and dietitian for the period of 8 weeks. Participants from the control group will receive general healthy eating recommendations.

We aim to investigate if the experiment had any effect on changes in metabolic, inflammation and nutritional markers, blood pressure and body weight and composition. Also, the effect of diets on men's sleep, general wellbeing and satisfaction with treatment will be investigated.

The proposed study can test a potentially effective nutritional intervention which is feasible to adopt and sustainable (in line with recent planetary diet recommendations). Confirming its effectiveness can fill the research gap, providing new knowledge and approach to the prevention and treatment of metabolic abnormalities in young, lean men.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 18-40 years
* Normal body weight
* At least one of metabolic abnormalities (elevated fasting glucose level - but not diabetes, elevated blood lipids, elevated blood pressure)

Exclusion Criteria:

* Females
* Age <18 and >40 years
* Overweight or obesity (BMI>25 kg/m2)
* WC > 94cm
* Alcohol >14 units/week
* Smoking
* On medication
* Diabetes or other chronic diseases
* Vegetarians or vegans
* Don't own or unable to use a Smartphone with Apple iOS or Android OS

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in glucose homeostasis | baseline, after 8 weeks and after 20 weeks from baseline
  Change in fasting glucose concentration [mg/dL]. Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas Integra 400 plus analyzer.

SECONDARY OUTCOMES:
Change in total cholesterol (TC) | baseline, after 8 weeks and after 20 weeks from baseline
  The blood serum concentration of total cholesterol (in mmol/L). Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas Integra 400 plus analyzer.
Change in high-density lipoprotein (HDL) cholesterol | baseline, after 8 weeks and after 20 weeks from baseline
  The blood serum concentration of high-density lipoprotein cholesterol (in mmol/L). Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas Integra 400 plus analyzer.
Change in low-density lipoprotein (LDL) cholesterol | baseline, after 8 weeks and after 20 weeks from baseline
  The blood serum concentration of low-density lipoprotein cholesterol (in mmol/L). Blood samples will be collected after the overnight fast and the analysis will be performed on Cobas Integra 400 plus analyzer.
Change in serum triglycerides (TG) | baseline, after 8 weeks and after 20 weeks from baseline
  The concentration of serum triglycerides (in mmol/L). Blood samples will be collected after the overnight fast and the analysis will be performed on Cobas Integra 400 plus analyzer.
Change in body weight | baseline, after 8 weeks and after 20 weeks from baseline
  Body weight (in kg) will be measured using a digital medical scale witl stadiometer.
Change in body mass index (BMI) | baseline, after 8 weeks and after 20 weeks from baseline
  The measured values of body height and weight will be used for the calculation of body mass index (in kg/m^2).
Change in body fat mass percentage | baseline, after 8 weeks and after 20 weeks from baseline
  Determination of body fat percentage will be performed using SECA® mBCA 515 analyser
Change in waist circumference | baseline, after 8 weeks and after 20 weeks from baseline
  Waist circumference measuring (in cm) will be performed using a non-strechable measuring tape.
Change in waist-to-hip ratio | baseline, after 8 weeks and after 20 weeks from baseline
  The waist-to-hip ratio will be calculated from the measured values of waist and hip circumferences: waist circumference (cm) / hip circumference (cm).
Change in visceral adipose tissue (VAT) | baseline, after 8 weeks and after 20 weeks from baseline
  Determination of abdominal fat volume will be measured in litres and performed using SECA® mBCA 515 analyser
Change in inflammatory markers-1 | baseline, after 8 weeks and after 20 weeks from baseline
  interleukin-6 [pg/mL] - COBAS e411 analyser
Change in inflammatory markers-2 | baseline, after 8 weeks and after 20 weeks from baseline
  C-reactive protein (CRP) [mg/L] - COBAS Integra 400 Plus analyser
Change in nutrition markers-1 | baseline, after 8 weeks and after 20 weeks from baseline
  Homocysteine [μmol/L] - COBAS Integra 400 Plus analyser
Change in nutrition markers-2 | baseline, after 8 weeks and after 20 weeks from baseline
  Vitamin B12 [pg/mL] - COBAS e411 analyser
Change in insulin concentration | baseline, after 8 weeks and after 20 weeks from baseline
  Insulin [units/mL] - COBAS e411 analyser
Change in haemoglobin glycosylated (HbA1c) concentration | baseline, after 8 weeks and after 20 weeks from baseline
  HbA1c [mmol/l] - COBAS e411 analyser
Change in systolic and diastolic blood pressure | baseline, after 8 weeks and after 20 weeks from baseline
  The assessment of blood pressure (in mmHg) will be performed prior to and immediately after the intervention using electronic monitor (Omron M3 Intellisense Automatic Blood Monitor, Omron Healthcare, Mannheim, Germany).

OTHER OUTCOMES:
Change in sleep length | baseline, after 8 weeks and after 20 weeks from baseline
  Measured using smartbands with sleep trackers: length (in hours)
Change in sleep quality | baseline, after 8 weeks and after 20 weeks from baseline
  Measured using smartbands with sleep trackers: with metrics specific to the selected model (score).
Change in cardiorespiratory fitness | baseline, after 8 weeks and after 20 weeks from baseline
  Oxygen consumption (VO2) measured using ergospirometer CORTEX MetaMax 3b (ml oxygen/kg of body weight/minute). VO2 max is the maximum amount of oxygen the body can utilize during exercise.
Change in physical activity level | baseline, after 8 weeks and after 20 weeks from baseline
  Measured using smartbands with pedometers (number of daily steps)
Participant's satisfaction with treatment upon completion | after 8 weeks
  Satisfaction with treatment: DSat-28 questionnaire (10.1002/osp4.299)
Change in dietary behaviours | baseline, after 8 weeks and after 20 weeks from baseline
  Dietary habits will be assessed using KomPAN questionnaire (https://doi.org/10.3390/nu10121845)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Lonnie, MSc, Principal Investigator — University of Warmia and Mazury in Olsztyn
Locations (1):
- University of Warmia and Mazury in Olsztyn, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: Undecided